CLINICAL TRIAL: NCT05109546
Title: Geriatric COVID-19 Serology
Acronym: SeroGerCov
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8438
Record Dates: First submitted 2021-11-04; First posted 2021-11-05 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Elderly people; Geriatric; RT-PCR SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronaviruses are important human and animal pathogens. At the end of 2019, a new coronavirus was identified as the cause of a cluster of pneumonia cases in Wuhan, a city in China's Hubei province. It quickly spread, leading to an epidemic across China, followed by an increasing number of cases in other countries around the world. In February 2020, the World Health Organization designated the disease COVID-19, which stands for coronavirus disease 2019. The virus that causes COVID-19 is SARS-CoV-2.

The duration of protection during which a patient after infection and / or vaccination remains clinically protected and the evolution of their serology as well as their titre remains unknown

ELIGIBILITY:
Inclusion criteria:

* Age> 75 years old
* Patient hospitalized or resident in the geriatrics center from July 1, 2020 to November 30, 2021 having presented with COVID or having benefited from a COVID vaccination.
* Subject not having expressed their opposition, after information, to the reuse of their data for the purposes of this research

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Impossibility of providing the subject with enlightened information (difficulties in understanding the subject, etc.)
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 76 Years | Sex: All
Age Groups: Older Adult
Study Population: Adult patient hospitalized or resident in the geriatrics center from July 1, 2020 to November 30, 2021 having presented with COVID or having benefited from a COVID vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of COVID serologies in a geriatric population after infection or vaccination | Files analysed retrospectively from July 1, 2020 to November 30, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Maxence MEYER, MD, Principal Investigator — Service SSR Gériatrique - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service SSR Gériatrique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France